CLINICAL TRIAL: NCT02689284
Title: A Phase 1b/2, Open Label, Dose Escalation Study of Margetuximab in Combination With Pembrolizumab in Patients With Relapsed/Refractory Advanced HER2+ Gastroesophageal Junction or Gastric Cancer
Brief Title: Combination Margetuximab and Pembrolizumab for Advanced, Metastatic HER2(+) Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGAH22-05
Record Dates: First submitted 2016-01-27; First posted 2016-02-23 (Estimated); Results first posted 2022-08-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Stomach Cancer; Esophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — margetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Margetuximab 10 mg/kg plus pembrolizumab 200 mg (Experimental): margetuximab administered in combination with pembrolizumab
  Interventions: Biological: Margetuximab 10 mg/kg; Biological: Pembrolizumab
- Cohort 2: Margetuximab 15 mg/kg plus pembrolizumab 200 mg (Experimental): margetuximab administered in combination with pembrolizumab
  Interventions: Biological: Margetuximab 15 mg; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Margetuximab 10 mg/kg — Margetuximab treatment is administered intravenously (IV) once every 21-day cycle
  Other Names: MGAH22
  Arms: Cohort 1: Margetuximab 10 mg/kg plus pembrolizumab 200 mg
Biological: Margetuximab 15 mg — Margetuximab treatment is administered IV once every 21-day cycle
  Other Names: MGAH22
  Arms: Cohort 2: Margetuximab 15 mg/kg plus pembrolizumab 200 mg
Biological: Pembrolizumab — Pembrolizumab treatment is administered IV once every 21-day cycle
  Other Names: MK-3475

SUMMARY:
This main purpose of this clinical study is to learn about the safety and activity of margetuximab and pembrolizumab combination treatment in patients with HER2+ gastric and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
Detailed Description: Both margetuximab and pembrolizumab are monoclonal antibodies used in combination to treat HER2+ gastric and gastroesophageal junction cancer. This study has two parts: Dose Escalation and Dose Expansion. The Dose Escalation phase of the study will evaluate safety of escalating doses of the combination treatment. The Dose Expansion phase will evaluate safety and activity of the combination in patients with gastric or gastroesophageal cancer once the final dose and schedule are defined. In addition, a cohort of patients with HER2+ 3+ gastric cancer patients will be enrolled in the Dose Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age ≥ 18 years old (or minimum age based upon local regulations)
3. Unresectable locally advanced or metastatic histologically proven HER2+ gastroesophageal junction (GEJ) or gastric cancer. Gastric Cancer Expansion Phase will include only gastric cancer patients with 3+ HER2 positivity.
4. HER2+ as 3+ (as defined in AJCC staging manual 8th edition) by IHC or in-situ hybridation (ISH) amplified.
5. Have received prior treatment with trastuzumab.
6. Have received treatment with at least one or more lines of cytotoxic chemotherapy in the metastatic setting.
7. Resolution of chemotherapy, immunotherapy or radiation-related toxicities.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Life expectancy ≥ 12 weeks.
10. Measurable disease as per RECIST 1.1 criteria.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) metastases.
2. Patients with any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, atopic dermatitis, or psoriasis not requiring systemic treatment.
3. History of prior allogeneic bone marrow, stem-cell or solid organ transplantation.
4. Treatment with any systemic anti-neoplastic therapy, or investigational therapy within the 3 weeks prior to the initiation of study drug.
5. Treatment with radiation therapy within 3 weeks prior to the initiation of study drug administration.
6. Treatment with corticosteroids (≥10 mg per day prednisone or equivalent) or other immune suppressive drugs within the 14 days prior to the initiation of study drug administration.
7. History of clinically-significant cardiovascular disease.
8. Clinically-significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation.
9. History of (non-infectious) pneumonitis that required steroids or presence of active pneumonitis
10. Clinically-significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis.
11. Evidence of active viral, bacterial, or systemic fungal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (11):
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute/Harvard University Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Swedish Cancer Institute, Seattle, Washington
- Canada (2):
  - Juravinski Cancer Centre - McMaster University, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Singapore (3):
  - National Cancer Centre, Singapore
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (9):
  - Kyungbuk National University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catenacci DV, Kang YK, Uronis HE, Lee KW, Ng MC, Enzinger PC, Park SH, Gold PJ, Lacy J, Hochster HS, Oh SC, Kim YH, Marrone KA, Kelly RJ, Juergens RA, Kim JG, Alcindor T, Sym SJ, Song EK, Chee CE, Chao Y, Kim S, Oh DY, Yen J, Odegaard JI, Lagow E, Li D, Sun J, Kaminker P, Moore PA, Rosales MK, Park H. Circulating Tumor DNA as a Predictive Biomarker for Clinical Outcomes With Margetuximab and Pembrolizumab in Pretreated HER2-Positive Gastric/ Gastroesophageal Adenocarcinoma. Oncology (Williston Park). 2023 Apr 25;37(4):176-183. doi: 10.46883/2023.25920992. PMID 37104758
- [Derived] Catenacci DVT, Kang YK, Park H, Uronis HE, Lee KW, Ng MCH, Enzinger PC, Park SH, Gold PJ, Lacy J, Hochster HS, Oh SC, Kim YH, Marrone KA, Kelly RJ, Juergens RA, Kim JG, Bendell JC, Alcindor T, Sym SJ, Song EK, Chee CE, Chao Y, Kim S, Lockhart AC, Knutson KL, Yen J, Franovic A, Nordstrom JL, Li D, Wigginton J, Davidson-Moncada JK, Rosales MK, Bang YJ; CP-MGAH22-5 Study Group. Margetuximab plus pembrolizumab in patients with previously treated, HER2-positive gastro-oesophageal adenocarcinoma (CP-MGAH22-05): a single-arm, phase 1b-2 trial. Lancet Oncol. 2020 Aug;21(8):1066-1076. doi: 10.1016/S1470-2045(20)30326-0. Epub 2020 Jul 9. PMID 32653053

RESULTS

PARTICIPANT FLOW:
Groups:
- Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg); Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg): combination treatment is administered once every 21-day cycle
Period: Overall Study
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Started | 3 | 92
Completed | 0 | 5
Not Completed | 3 | 87
Not completed — Adverse Event | 1 | 8
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — progression of cancer | 1 | 72
Not completed — decreased heart function | 0 | 1
Not completed — concern for anemia | 0 | 1
Not completed — no measurable cancer for evaluation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg) | Total
Number analyzed (Participants) | 3 | 92 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.87) | 60.2 (12.83) | 60.3 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 17 | 17
  Male | 3 | 75 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 88 | 91
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 51 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 3 | 34 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 3 | 3
  South Korea | 0 | 42 | 42
  Singapore | 0 | 8 | 8
  United States | 3 | 38 | 41
  Taiwan | 0 | 1 | 1
ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status is a 0-5 measurement of the participant's limitations on everyday activities due to cancer. A score of 0 indicates fully active; no performance restrictions. A score of 1 indicates strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  participants
    0 | 0 | 33 | 33
    1 | 3 | 59 | 62
Primary tumor location [Number; unit: participants]
  Gastric | 0 | 61 | 61
  Gastroesophageal junction | 3 | 31 | 34
HER2 status using immunohistochemistry (IHC) [Count of Participants; unit: Participants] — HER2 is a growth factor present in some gastric cancers HER2 stats is a measure of how much HER2 is present in the cancer tissue and how sensitive the cancer may be to HER2 blockage. Participants with cancer that is IHC 3+ are most sensitive to treatment with a HER2 inhibitor like margetuximab.
  Participants
    IHC 2+ | 2 | 21 | 23
    IHC 3+ | 1 | 71 | 72
PD-L1 Status [Count of Participants; unit: Participants] — PD-L1 is present in some gastric cancers. Participants with cancer that is PD-L1+ are most sensitive to treatment with immunotherapy like pembrolizumab.
  Participants
    PD-L1 positive | 1 | 33 | 34
    PD-L1 negative | 1 | 43 | 44
    unknown | 1 | 16 | 17
HER2 IHC 3+ and PD-L1 positive [Count of Participants; unit: Participants] | 0 | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities
Description: Characterize maximum tolerated dose (MTD) or maximum administered dose (MAD) (if no MTD is defined) of margetuximab when administered in combination with pembrolizumab
Time Frame: 21 days
Population: Dose escalation cohorts to determine the expansion cohort dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Number of Patients With Adverse Events (AEs) and Serious Adverse Events (SAEs).
Description: The number of patients that experience either an AE or a SAE during the study participation
Time Frame: up to 24 months
Population: All patients receiving at least 1 dose of margetuximab or pembrolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
Participants | 3 | 86

3. Primary Outcome: Number of Patients With a Complete Response (CR) or Partial Response (PR) to Treatment
Description: Investigate the preliminary anti-tumor activity as measured by response to treatment of margetuximab when administered in combination with pembrolizumab, using conventional Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
Participants | 0 | 18

4. Primary Outcome: Number of Patients With a Complete Response (CR) or Partial Response (PR) to Treatment Using irRC Criteria
Description: Investigate the preliminary anti-tumor activity, as measured by objective response rate (ORR) of margetuximab when administered in combination with pembrolizumab, using immune-related response criteria (irRC).
Time Frame: 12 Months
Population: Analysis is limited to patients receiving margetuximab (15 mg/kg) and pembrolizumab (200 mg)
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
Participants | 0 | 19

5. Primary Outcome: Duration of Response
Description: Duration of response is calculated at the time from CR or PR to relapse or cancer progression.
Time Frame: up to 24 months
Population: There were no responders in the 10mg/kg group
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 0 | 92
months |  | 12.1 [2.79 to 26.68]

6. Secondary Outcome: Overall Survival (OS)
Description: The median length of time between first dose of study medication and death from any cause.
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
months | 7.0 [2.37 to 9.66] | 12.7 [9.07 to 14.62]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: The interval between the first dose of study medication and progression of disease or death from any cause.
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
months | 1.4 [1.31 to 2.76] | 2.7 [0.37 to 4.34]

8. Secondary Outcome: Change From Baseline in Pharmacodynamic Markers in Whole Blood
Description: The planned assessment included examination of markers of T-cell activation
Time Frame: from first dose to the end of treatment, average about 12 months
Population: Analysis was not performed. A number of samples were degraded in shipping rendering insufficient samples to conduct the analysis.
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Analysis of HER2 Tumor Cell Membrane Expression in Biopsy Specimens Before and After Treatment
Time Frame: from first dose to the end of treatment, average 12 months.
Population: Sample collection was planned for the Margetuximab (15 mg/kg) plus pembrolizumab (200 mg) cohort only. No samples were received that could be tested. The analysis could not be conducted.
Arm/Group | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Patients Who Develop Treatment-emergent Anti-drug Antibodies to Margetuximab (Immunogenicity)
Time Frame: Assessed Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Day 1 of every odd cycle, and end of treatment visit, average 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
Participants | 1 | 4

11. Secondary Outcome: Maximum Concentration of Margetuximab at Steady State
Description: Measurement of PK characteristics is limited to margetuximab. No analysis of pembrolizumab was conducted.
Time Frame: At end of infusion on Cycle 1, Day 1. Cycle 2, Day 1; Cycle 3, Days 1 and 2; Cycle 5 Day 1, Cycle 7 Day 1, and end of treatment visit, average 12 months
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
mcg/mL | 197 (0.249) | 318 (0.168)

12. Secondary Outcome: Area Under the Concentration Time Curve at Steady State (AUC ss)
Description: AUC is a mathematical calculation that describes the variation in drug concentration in the blood over time.
Time Frame: Predose and at end of infusion on Cycle 1, Days 1, 2 and 8: Cycle 2, Day 1; Cycle 3, Days 1 and 2; Cycle 5 Day 1, Cycle 7 Day 1, and end of treatment visit, average 12 months
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL* day
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
mcg/mL* day | 1710 (0.358) | 2720 (0.329)

13. Secondary Outcome: Clearance
Description: Drug clearance is the amount of drug removed from the bloodstream by the body per unit of time.
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per day
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
liters per day | 0.381 (0.0394) | 0.329 (0.296)

14. Secondary Outcome: Volume of Distribution at Steady State
Description: The volume of distribution is related to a whether how much drug is distributed to body tissues, or remains in the bloodstream.
Time Frame: Predose and at end of infusion on Cycle 1, Days 1, 2 and 8: Cycle 2, Day 1; Cycle 3, Days 1 and 2; Cycle 5 Day 1, Cycle 7 Day 1, and end of treatment visit average 12 months .
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
liters | 7.7 (0.306) | 6.37 (0.205)

15. Secondary Outcome: Terminal Half-life
Description: Terminal half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Time Frame: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
Number analyzed (Participants) | 3 | 92
day | 17.2 (0.312) | 16.2 (0.286)

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the time of first dose through 28 days after the last dose or until the start of another anti-cancer treatment, whichever was earlier, average 12 months.
Description: Adverse event reporting is based on physical examination findings, patient reports, and clinically significant abnormal laboratory values.
  Progression of the underlying neoplasm resulting in hospitalization or death was documented as an antitumor activity outcome and not as an SAE, unless considered drug-related by the investigator. If an SAE occured in a patient and it was unclear whether the event was related to progressive disease, the SAE was reported.
Arm/Group | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg)
All-Cause Mortality (participants affected / at risk) | 3/3 | 69/92
Serious Adverse Events (participants affected / at risk) | 2/3 | 38/92
Other Adverse Events (participants affected / at risk) | 3/3 | 86/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) (N=3) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg) (N=92)
Anaemia (Blood and lymphatic system disorders) | 0 | 9
Hypophysitis (Endocrine disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 2
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2
Eye infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Adnexal torsion (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab (10 mg/kg) Plus Pembrolizumab (200 mg) (N=3) | Margetuximab (15 mg/kg) Plus Pembrolizumab (200 mg) (N=92)
Anaemia (Blood and lymphatic system disorders) | 0 | 29
Diarrhoea (Gastrointestinal disorders) | 1 | 26
Nausea (Gastrointestinal disorders) | 0 | 23
Abdominal pain (Gastrointestinal disorders) | 0 | 16
Vomiting (Gastrointestinal disorders) | 0 | 16
Dyspepsia (Gastrointestinal disorders) | 0 | 12
Constipation (Gastrointestinal disorders) | 1 | 10
Dysphagia (Gastrointestinal disorders) | 0 | 8
Abdominal distension (Gastrointestinal disorders) | 0 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6
Fatigue (General disorders) | 1 | 25
Oedema peripheral (General disorders) | 0 | 10
Pyrexia (General disorders) | 0 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 12
Weight decreased (Investigations) | 0 | 11
Amylase increased (Investigations) | 0 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 6
Lipase increased (Investigations) | 0 | 6
Alanine aminotransferase increased (Investigations) | 0 | 5
Blood creatinine increased (Investigations) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Dizziness (Nervous system disorders) | 0 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 5
Insomnia (Psychiatric disorders) | 0 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 18
Rash (Skin and subcutaneous tissue disorders) | 0 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT02689284/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02689284/SAP_001.pdf